| Official Title: | Modifying Young Adult Skin Cancer Risk and Protective Behaviors |
|---|---|
| NCT number: | NCT03313492 |
| <b>Document Type:</b> | Consent Form: Main |
| Date of the | 08/02/2018 |
| Document: | |

### Informed Consent Form

Study Title: Young Adult Skin Cancer Risk and Protective Behaviors
UV4.me2

You are being asked to participate in a research study that is being conducted by the at . This is a study on skin cancer prevention that is being conducted by .

#### Purpose of the study:

This is a research study. Research studies include only people who choose to take part. If you have any questions, you can contact us for more information. You are being asked to take part in this research study because you are a young adult at moderate to high risk of getting skin cancer, based on the screening questions you answered.

The sponsor of this study is the

Skin cancer is the most common cancer, and it can be deadly. Ultraviolet (UV) rays can also affect your looks and health in other ways. The purpose of this study is to learn how to help young adults reduce their risk for skin cancer. You will be one of approximately 1,500 study participants.

#### What will happen?

In this study, you will fill out online questionnaires and view online material about skin protection, UV rays, and skin cancer. Many people find the questionnaires and material interesting and fun.

#### Questionnaires

We are asking you to fill out questionnaires for this research study. These questionnaires will tell us about your background, skin protection and risk behaviors and attitudes, and opinions of the study. You will spend about 10 minutes filling out each of the questionnaires. We will ask you to fill them out five times during this research study.

## Randomization

You will be "randomized" into one of three research study groups. Randomization means that you are put into a group by chance. A computer program will place you in one of the research study groups. Neither you nor the study team can choose the group you will be in. Each of the three study groups involves taking questionnaires and viewing a different type of skin cancer prevention material online.

How long will you be in the research study? You will be in this study for about 12 months.

# Participation

Participation in this study is voluntary. The only alternative to this study is not to participate.

# Risks or discomforts:

Possible risks related to the study include: the time and effort it takes to complete the study, slight distress when considering health risks, and/or breach of confidentiality. We will do our best to lessen these risks as much as possible and help you with them if they happen. You may withdraw from the study at any time. If you decide to quit before you have finished a questionnaire, your answers will NOT be recorded.

The study may involve risks which are currently unforeseeable. You should talk to the study representative about any problems that you have while taking part in the research study.

APPROVE IRB ID:
Approval Date:
Expiration Date:

#### Benefits of this study:

We hope that you will enjoy the study and find it interesting and fun. You may learn about how to protect your skin and decrease your risk of skin cancer. You will also assist us in learning how to help other people prevent skin cancer. It is possible that the study will not benefit you directly.

#### Confidentiality:

The researchers will see your individual questionnaire responses and the activities you complete within the website. We ask you to include your name, email address, and phone number so that we can remind you from time to time about the questionnaires and the skin cancer prevention program by email and/or text. If we receive your questionnaires on time, it is unlikely that we would try to call you. You will be assigned a participant number. Data are encrypted. Once data collection is complete, your contact information will be deleted, and no link between the questionnaire data and your identity will exist.

We will do our best to make sure any personal information you give us will be kept private. However, we cannot guarantee total privacy. Your personal information may be given out if required by law. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used. Organizations that may look at and/or copy your responses for research, quality assurance, and data analysis include:

and its affiliates or subsidiaries and other authorized representatives of these organizations.

This research is covered by a Certificate of with this Certificate may not disclose or use information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below). The Certificate cannot be used to refuse a request for information from personnel of the United States federal or state government agency sponsoring the project that is needed for auditing or program evaluation by this project or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). You should understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

#### Compensation:

If you complete the study activities as instructed, you will be eligible to receive an electronic gift-card for filling out a questionnaire at the following time-points: 1 month = \$10, 3 months = \$15, 6 months = \$20, and 12 months = \$25. You will also receive \$5 for completing the baseline questionnaire and viewing the skin cancer prevention material for the first time plus a \$25 bonus if you complete all five questionnaires, for a possible total of \$100 throughout the year. You may choose to be entered in a raffle for \$100 at each of the five time-points. In one of the groups, you will also be able to earn discounts for skin care products such as sunscreen and protective clothing and eyewear. We will not share any information about you or your study participation with the companies providing these discounts.

#### Withdrawal:

Your participation is voluntary; you are free to withdraw your participation from this study at any time. If you do not want to continue, you can simply leave the website or let us know. If you do not click on a "submit" button at the end of the questionnaire, your answers and participation will not be recorded. Research staff may stop you from taking part in the study if you do not follow the study rules.

## How the findings will be used:

The results of the study will be used for research. The results from the study will be presented at academic and/or professional conferences, and the results might be published in an academic or professional journal.

#### Contact information:

2 Version #:2 7/26/18



| clicking this box and typing your name, you acknow participate in this research, with the knowledge that you lif you do not wish to take part in this study, exit this page study later if you prefer. | |
|---|---|
| First Name | Last Name |
| You can print a copy of this form for your records. So that please give a secondary email address and phone number. | we can reach you during the study only if necessary,<br>You can ask us to stop contacting you at any time. |
| Secondary Email Address (optional) | Secondary Phone Number (optional) |
| ACCEPT AND CONTINUE | |

